CLINICAL TRIAL: NCT03065933
Title: An Extended-Release Form of Clonidine as an Anti-Manic Agent: An Add-On, Open-Label Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth S. Liebson, PI, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-P-002018/1; McLean
Record Dates: First submitted 2012-11-06; First posted 2017-02-28 (Actual); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Bipolar Disorder, Mania
Keywords: mania; clonidine; bipolar disorder
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Clonidine

STUDY DESIGN:
Intervention Model Description: Subjects with Bipolar Disorder, mania will receive an extended-release from of clonidine on the second day of this 3-day study. Rating scale, record of sleep, and a questionnaire of adverse effects will be recorded on each of the 3 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- clonidine as an antimanic agent (Experimental): Subjects with Bipolar Disorder, Mania receive an extended-release form of clonidine on the second day of this 3-day study. Rating scales, record of sleep, and a questionnaire of adverse effects is recorded on each of the three days.
  Interventions: Drug: extended-release clonidine

INTERVENTIONS:
Drug: extended-release clonidine — Subjects will received 0.2 mg extended-release clonidine twice on second day of this three-day study.
  Other Names: Kapvay

SUMMARY:
The investigators plan to to study an extended-release form of clonidine, which the investigators hope will be even better tolerated than the immediate-release form, as an antimanic agent. Subjects will receive an extended-release form of clonidine in addition to their usual medication regimen on the second day of this three-day study. Rating scales, a record of sleep, and a questionnaire of adverse effects will be recorded on each of the 3 days. Any medication changes made by the attending psychiatrist and prns administered will be recorded throughout the study.

DETAILED DESCRIPTION:
Clonidine has been reported to be effective in a variety of hyperadrenergic states, including mania. It is generally well-tolerated and does not result in the severe adverse effects that are associated with many antipsychotics and mood stabilizers used in the treatment of mania, such as weight gain and akathisia. There is some suggestion that clonidine may be particularly effective in a subset of refractory cases and in patients who cannot tolerate antipsychotic medications or lithium. The investigators plan to to study an extended-release form of clonidine, which the investigators hope will be even better tolerated than the immediate-release form, as an antimanic agent. Subjects will receive an extended-release form of clonidine in addition to their usual medication regimen on the second day of this three-day study. Rating scales, a record of sleep, and a questionnaire of adverse effects will be recorded on each of the 3 days. Any medication changes made by the attending psychiatrist and prns administered will be recorded throughout the study. The investigators believe that studying as few as 10 subjects will give the investigators a sense as to whether the addition of clonidine is helpful in reducing manic symptoms and if the rate of adverse effects is unacceptable.

ELIGIBILITY:
Inclusion Criteria:

* meet SCID criteria for bipolar disorder, type I, Mania with YMRS > 15
* No significant improvement in symptoms after three or more days of hospitalization
* documented medical evaluation without identified acute or serious medical illness
* negative pregnancy test in women of child-bearing age

Exclusion Criteria:

* involuntary commitment or lack of capacity to provide informed consent
* low blood pressure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Cohen, MD, PhD, Study Chair — Mclean Hospital

IPD SHARING:
Plan to Share IPD: Yes
IPD to be shared via clinicaltrials.gov, publication, or personal request.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clonidine as an Antimanic Agent
Started | 5
Completed | 0
Not Completed | 5
Not completed — study terminated | 5

BASELINE CHARACTERISTICS:
Population: No data besides region of enrollment was collected on these participants before the study terminated.
Arm/Group | Clonidine as an Antimanic Agent
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: No data was collected on the 5 participants, except for region of enrollment, before the study terminated.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: No data was collected on the 5 participants, except for region of enrollment, before the study terminated.
Region of Enrollment [Count of Participants; unit: Participants] — Population: All participants were enrolled in the United States, but no other data was collected.
  Participants
    United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Score on a Mania Rating Scale
Description: Mania rating scale to be performed each day of this 3 day study.
Time Frame: 3 days
Population: No data was collected on the 5 participants, except for region of enrollment, before the study terminated.
Arm/Group | Clonidine as an Antimanic Agent
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: No data was collected on the 5 participants enrolled, except for region of enrollment, before the study terminated.
Arm/Group | Clonidine as an Antimanic Agent
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes